CLINICAL TRIAL: NCT01069588
Title: ACL Reconstruction - Bioabsorbable Screws- 2 Year Follow-up
Brief Title: Anterior Cruciate Ligament (ACL) Reconstruction- Bioabsorbable Screw
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Kurt P. Spindler, Professor, Vanderbilt University Medical Center
Other Study IDs: 090805
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: bioabsorbable screw; acl reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Calaxo: Received Calaxo screw
- Milagro: Received a Milagro screw

SUMMARY:
To evaluate the knee functionality, screw integrity, graft integrity, cartilage effect, and bony ingrowth in patients treated with the CALAXO screw and MILAGRO screw two years after ACL reconstruction.

DETAILED DESCRIPTION:
This study will combine the use of survey response, MRI, and x-rays of the knees in Dr. Spindler's ACL reconstructed patients in order to examine long term healing of two types of bioabsorbable screw. We will use a 2-4 yr time point to look at patient reported symptoms of pain and swelling from the surveys and use the x-rays and MRIs to look at absorption of the screw, healing of the graft, and body reactions to the screw.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 12-35 years of age at the time of follow-up.
* Gender: Both.
* Minorities: All.
* Involved in sports at the time of injury.
* Participants must be at least two years past the date of ACL reconstruction surgery and not more than four years past the date of surgery
* Bioabsorbable Screws used during ACL reconstruction surgery

Exclusion Criteria:

* Age: <12 or >35 years of age
* Non-active or unable to participate for health reasons
* Simultaneous bilateral ACL reconstruction surgeries.
* If any of the following conditions exist in the ipsilateral knee:

  * Revision ACL reconstruction
  * Complex knee injury
* If any of the following conditions exist in the contralateral knee:

  * ACL deficient
  * Prior ACL reconstruction
  * Prior surgery of any type
* Insufficient initial documentation
* Cannot be contacted by phone
* Neither Calaxo nor Milagro screw used at the time of ACL reconstruction

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 2-4 years post ACL reconstruction performed by Dr. Kurt Spindler, under age 35, injured in sport, unilateral primary ACL.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Screw integrity | 2-4 yrs
Tunnel enlargement | 2-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurt P Spindler, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Cox CL, Spindler KP, Leonard JP, Morris BJ, Dunn WR, Reinke EK. Do newer-generation bioabsorbable screws become incorporated into bone at two years after ACL reconstruction with patellar tendon graft?: A cohort study. J Bone Joint Surg Am. 2014 Feb 5;96(3):244-50. doi: 10.2106/JBJS.L.01652. PMID 24500587